CLINICAL TRIAL: NCT05507294
Title: A Clinical Study to Evaluate Food Effect on Pharmacokinetics and Safety After Single Dose Glumetinib in Healthy Chinese Male Subjects
Brief Title: Single Dose Glumetinib in Healthy Chinese Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Haihe Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: SCC244-106
Record Dates: First submitted 2022-08-17; First posted 2022-08-18 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Healthy Volunteers
Keywords: Healthy Chinese Male Subjects; SCC244; Food effect
MeSH Terms: interventions — glumetinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- SCC244：Fasting+High-fat meal+Low-fat meal (Experimental): Participants will receive a single oral dose of Glumetinib tablet in fasting condition on Day 1 of treatment period 1 followed by a single oral dose of Glumetinib tablet in fed condition(High-fat meal) on Day 1 of treatment period 2.Then，Participants will receive a single oral dose of Glumetinib tablet in fed condition （Low-fat meal）on Day 1 of treatment period 3. The time interval between two adjacent dosages was at least 14 days.
  Interventions: Drug: Glumetinib
- SCC244：Fasting+Low-fat meal+High-fat meal (Experimental): Participants will receive a single oral dose of Glumetinib tablet in fasting condition on Day 1 of treatment period 1 followed by a single oral dose of Glumetinib tablet in fed condition(Low-fat meal) on Day 1 of treatment period 2.Then，Participants will receive a single oral dose of Glumetinib tablet in fed condition （High-fat meal）on Day 1 of treatment period 3. The time interval between two adjacent dosages was at least 14 days.
  Interventions: Drug: Glumetinib
- SCC244：High-fat meal+Fasting+Low-fat meal (Experimental): Participants will receive a single oral dose of Glumetinib tablet in fed condition（High-fat meal） on Day 1 of treatment period 1 followed by a single oral dose of Glumetinib tablet in fasting condition on Day 1 of treatment period 2.Then，Participants will receive a single oral dose of Glumetinib tablet in fed condition(Low-fat meal) on Day 1 of treatment period 3. The time interval between two adjacent dosages was at least 14 days.
  Interventions: Drug: Glumetinib
- SCC244：High-fat meal+Low-fat meal+Fasting (Experimental): Participants will receive a single oral dose of Glumetinib tablet in fed condition（High-fat meal） on Day 1 of treatment period 1 followed by a single oral dose of Glumetinib tablet in fed condition（Low-fat meal） on Day 1 of treatment period 2.Then，Participants will receive a single oral dose of Glumetinib tablet in fasting condition on Day 1 of treatment period 3. The time interval between two adjacent dosages was at least 14 days.
  Interventions: Drug: Glumetinib
- SCC244：Low-fat meal+Fasting+ High-fat meal (Experimental): Participants will receive a single oral dose of Glumetinib tablet in fed condition（Low-fat meal） on Day 1 of treatment period 1 followed by a single oral dose of Glumetinib tablet in fasting condition on Day 1 of treatment period 2.Then，Participants will receive a single oral dose of Glumetinib tablet in fed condition(High-fat meal) on Day 1 of treatment period 3. The time interval between two adjacent dosages was at least 14 days.
  Interventions: Drug: Glumetinib
- SCC244：Low-fat meal +High-fat meal +Fasting (Experimental): Participants will receive a single oral dose of Glumetinib tablet in fed condition（Low-fat meal） on Day 1 of treatment period 1 followed by a single oral dose of Glumetinib tablet in fed condition（High-fat meal） on Day 1 of treatment period 2.Then，Participants will receive a single oral dose of Glumetinib tablet in fasting condition on Day 1 of treatment period 3. The time interval between two adjacent dosages was at least 14 days.
  Interventions: Drug: Glumetinib

INTERVENTIONS:
Drug: Glumetinib — Fasting: Subjects are fasted overnight (at least 10 hours before administration) and receive Glumetinib tablets with 240 mL warm water the next morning.
  Fed (high-fat meal/low-fat meal): Following an overnight fast for at least 10 hours, subjects finished a high-fat meal, or a low-fat meal within 30 minutes the next morning (eat up all meals). Glumetinib tablets are orally administered by subjects with 240 mL warm water on 30 minutes after starting the meal. Water is allowed as desired except for 1 hour before and 2 hours after administration (including the meal), and no more than 500 mL of water will be consumed including the water intake during the high-fat meals or low-fat meals, and the water for administration. The subjects will be fasted for at least 4 hours after administration, and then have dinner approximately 9 hours after administration.
  Other Names: SCC244

SUMMARY:
This is a phase I, single-center, randomized, open-label, single-dose, three-period (fasting, high-fat meal, low-fat meal) crossover clinical study to investigate the food effect on PK of the recommended phase II dose (RP2D) of 300 mg Glumetinib, based on the previous clinical studies of Glumetinib monotherapy.

DETAILED DESCRIPTION:
Approximately 18 healthy adult male subjects are expected to be enrolled randomly into 6 meal sequences, with 3 subjects per sequence. Each subject receive Glumetinib given under fasting condition, after a high-fat meal, or following a low-fat meal, respectively, in three periods.Subjects enrolled in each period received 300 mg Glumetinib once and PK blood samples are collected after dosing once daily for 7 days.To clarify the occurrence of AEs, subjects should complete safety examinations on Day 8 of each period. Subjects with AE are followed up before the next period of administration. Before the next administration, subjects with no AE or ongoing AE with Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 enter into the next period and continued receiving dosing; subjects reported AEs with CTCAE Grade higher than 1 are discontinued from the study and are followed up by investigator until the AE disappeared, stabilized, return to baseline or lost to follow-up (whichever occurred first)

ELIGIBILITY:
Inclusion Criteria:

* Subjects has to meet all of the following criteria for study entry:

  1. Healthy Chinese male subjects are 18 to 45 years of age, inclusive. "Healthy" in this criterion refers to normal results of medical history interview, physical examinations, vital sign measurements, clinical laboratory tests, chest X-ray (posteroanterior [PA]) and 12-lead electrocardiogram (ECGs), or abnormalities with no clinical significance as judged by the investigator.
  2. Bodyweight ≥50.0 kg and body mass index (BMI) are between 19.00 and 26.00 kg/m2, inclusive.
  3. Subjects should be able to take adequate and effective contraceptive measures and to avoid sperm donation during the study (from the informed consent form [ICF] signed to the last visit completed), and within 6 months after the end of the study.

     Adequate and effective contraception is defined as the following:
     * Complete abstinence: If it is consistent with subject's preference or lifestyle.
     * Adhere to the correct use of one of the following birth control measures:

       1. Use of an intra-uterine device (IUD) by the subject's female partner; or
       2. Barrier measures such as diaphragm or condom.
  4. Subjects should sign the ICF voluntarily and understand the purpose, process and risks of the study.
  5. Subjects should be able to communicate well with the investigator and comply with the requirements of the clinical study.

Exclusion Criteria:

* Subjects who has any of the following diseases or conditions

  1. Known malignancy or psychiatric disorder.
  2. Known to suffer from acute/chronic bronchospasm (asthma, chronic obstructive pulmonary disease, etc.), pulmonary fibrosis, pulmonary tuberculosis and other diseases that affect respiratory function.
  3. Has a history of diabetes mellitus and/or pancreatitis.
  4. History of major gastrointestinal surgery (except appendicitis surgery, anal prolapse surgery), such as gastrectomy, gastroenterostomy, enterectomy, gastric bypass, gastric division or gastric banding, etc.
  5. Headache ≥2 per week and duration ≥30 minutes within 3 months, or headache episode within 1 week before administration.

     Subjects who has any of the following diseases or clinically significant abnormalities at the screening examination
  6. Suffering from allergic diseases (such as allergic rhinitis, allergic asthma), had a history of systemic allergic reactions, allergies to any component of the study drug or allergies to similar drugs
  7. Uncured pulmonitis, blood system, respiratory system, cardiovascular and cerebrovascular system, and digestive system disorders with clinical significance, and any known diseases that may affect drug absorption, distribution, metabolism and excretion.
  8. Mean corrected QT interval (QTcF) at rest > 450 ms by 12-lead ECG, or other abnormalities with clinical significance in the opinion of the investigator.
  9. Positive results for hepatitis B virus surface antigen (HBsAg), anti-hepatitis C virus (HCV) antibody, treponema pallidum antibody; and non-negative for human immunodeficiency virus (HIV) antibody.

     Subjects who has any of the following conditions within a certain period before the screening/baseline (i.e., the day before the first period of administration, D-1) examination
  10. Consumed foods that affect the liver drug enzyme CYP3A4 (such as grapefruit or beverages containing grapefruit) or foods or beverages rich in xanthine (such as chocolate, coffee, red bull, etc.) within 48 hours before administration.
  11. Use any over-the-counter drugs (including vitamins and herbal supplements, etc., except vitamin-containing beverages) within one week.
  12. Use of any prescription drug within 2 weeks or less than 5 half-lives between the last prescription drug and the first dose of Glumetinib, whichever is shorter.
  13. Smoking ≥5 cigarettes per day within 3 months or unable to refrain from smoking during the study.
  14. Regular drinkers (exceeding 2 units of alcohol per day on average [1 unit = 360 mL beer or 45 mL spirits with 40% alcohol or 150 mL wine]) within 3 months or a positive alcohol breath test at screening/baseline.
  15. History of drug abuse within 12 months before screening examination or positive urine drug abuse screening test during the screening/baseline.
  16. Blood donation or blood loss ≥300 mL within 3 months.
  17. Participation in any other clinical studies (including clinical studies of drugs and medical devices) within 3 months.
  18. Other conditions that the investigator considered inappropriate for the subject to participate in the clinical trial.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 18 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2021-05-21 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
AUC0-inf | Blood samples are collected pre-dose, 0.5, 1, 2, 2.5,3, 3.5,4, 6, 8, 12, 24,36, 48, 72, 96,120, 168 hours post dose)
  Area Under the Concentration-time Curve from Time zero to Infinity
AUC0-t | Blood samples are collected pre-dose, 0.5, 1, 2, 2.5,3, 3.5,4, 6, 8, 12, 24,36, 48, 72, 96,120, 168 hours post dose
  Area Under the Concentration-Time Curve from Time Zero to Last Measurable Time Point
Cmax | Blood samples are collected pre-dose, 0.5, 1, 2, 2.5,3, 3.5,4, 6, 8, 12, 24,36, 48, 72, 96,120, 168 hours post dose
  Maximum Plasma Concentration
Tmax | Blood samples are collected pre-dose, 0.5, 1, 2, 2.5,3, 3.5,4, 6, 8, 12, 24,36, 48, 72, 96,120, 168 hours post dose
  Time at Maximum Plasma Concentration (Cmax)
t1/2 | Blood samples are collected pre-dose, 0.5, 1, 2, 2.5,3, 3.5,4, 6, 8, 12, 24,36, 48, 72, 96,120, 168 hours post dose
  Half-Life
CL/F | Blood samples are collected pre-dose, 0.5, 1, 2, 2.5,3, 3.5,4, 6, 8, 12, 24,36, 48, 72, 96,120, 168 hours post dose
  Apparent Clearance
V/F | Blood samples are collected pre-dose, 0.5, 1, 2, 2.5,3, 3.5,4, 6, 8, 12, 24,36, 48, 72, 96,120, 168 hours post dose
  Apparent Volume of Distribution

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hositpal, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No